CLINICAL TRIAL: NCT04671238
Title: Absolute Quantification in Bone Scintigraphy: Phantom Evaluation and Clinical Application in Patients Undergoing Follow-up for Vertebral Fractures.
Brief Title: Absolute Quantification in Bone Scintigraphy
Acronym: QUANTOSS-3D
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre Yves MARIE, Study director, Central Hospital, Nancy, France
Other Study IDs: 2020PI241
Record Dates: First submitted 2020-11-13; First posted 2020-12-17 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Scintigraphy Quantification
Keywords: bone scintigraphy; absolute quantification; Standard Uptake Value
MeSH Terms: interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient for SPECT/CT scan: Patients referred for SPECT/CT scan of the spine as part of a vertebroplasty workup and selected retrospectively.
  Interventions: Device: SPECT CT

INTERVENTIONS:
Device: SPECT CT — SPECT/CT scan of the spine as part of a vertebroplasty

SUMMARY:
While absolute quantification in 18F-FDG PET (Positon Emission Tomography) is widely used in clinical routine, absolute quantification in SPECT (Single Photon Emission Computed Tomography) is under development and its clinical interest remains to be demonstrated. Recent studies carried out on bone scan recordings show the potential interest of quantification indexes such as SUV (Standard Uptake Value).

DETAILED DESCRIPTION:
In oncology, bone scan studies have reported significantly higher SUV values for secondary bone lesions compared with benign osteoarticular lesions , and some have even defined an SUVmax threshold value that points to prostatic bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent vertebral fractures:

  1. who have had at least two SPECT/CT scan scans of the spine as part of a pre-vertebroplasty check-up,
  2. for which fracture dates were known.

Exclusion Criteria:

1. Minor person
2. Person opposing the use of their data (Posters in waiting rooms explaining that the patient must object if they do not wish their data to be used)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for SPECT/CT scan of the spine as part of a vertebroplasty workup and selected retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
To validate the absolute bone scan quantification in a retrospectively selected patient population | After 1 year
  Analysis of SUV variation on at least 2 bone scans: Variation of the SUV over time on scans of patients with spinal fractures

SECONDARY OUTCOMES:
To calibrate the tomographic images from the gamma camera | 1 day
  Calibrate the tomographic images from the gamma camera to obtain a volume activity in Bq/mLand densities
To evaluate the attenuation correction on phantoms of different density | 1 day
  SUV absolute quantitation index (SUVmax, SUVpeak, SUVmean).
To evaluate absolute quantification on phantoms | 1 day
  Evaluate absolute quantification on phantoms with objects of different volumes

CONTACTS AND LOCATIONS:
Overall Officials: BALHOUL Achraf, MD, Principal Investigator — CHRU of Nancy
Locations (3):
- France (3):
  - CHU de Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
  - Chru Nancy, Vandœuvre-lès-Nancy
  - CHRU of Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No